CLINICAL TRIAL: NCT00310219
Title: Comparative Study of Gross Tumor Volume Definition With or Without PET Fusion for Patients With Non-Small Cell Lung Carcinoma
Brief Title: Positron Emission Tomography Scan and CT Scan in Planning Radiation Therapy for Patients With Stage II or Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RTOG-0515; CDR0000465501
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Two radiation oncologists are randomly assigned to develop either a 3DCRT plan using CT only, or a 3DCRT plan using fused PET/CT
  Interventions: Procedure: computed tomography; Procedure: positron emission tomography

INTERVENTIONS:
Procedure: computed tomography
Procedure: positron emission tomography

SUMMARY:
RATIONALE: Imaging procedures, such as positron emission tomography (PET) scan and CT scan, may help doctors plan radiation therapy for patients with non-small cell lung cancer.

PURPOSE: This clinical trial is studying how well a combined PET scan and CT scan works compared to a CT scan alone in planning radiation therapy for patients with stage II or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the impact of positron emission tomography (PET)/CT fusion scan and CT scan alone, by comparing gross tumor volume (GTV) contours and three-dimensional conformal radiotherapy treatment plans using 2 separate data sets (PET/CT fusion scan and CT scan only), in patients with stage II or III non-small cell lung cancer who are planning to undergo radiotherapy.
* Determine the impact of PET on GTV (cm^3), number of involved nodes, location of involved nodes, and dosimetric measures of normal tissue toxicity (mean lung dose, V20, and mean esophageal dose).

Secondary

* Determine the rate of elective nodal failures (nodal failures in regions that are not intentionally irradiated to definitive doses [i.e., ipsilateral hilum, mediastinum, or ipsilateral supraclavicular fossa]).

OUTLINE: This is a multicenter study. Patients are stratified according to neoadjuvant chemotherapy (yes vs no).

Patients undergo a combined positron emission tomography (PET)/CT scan. Patients also undergo a CT scan alone. A single three-dimensional conformal radiotherapy (3DCRT) plan is generated from the combined PET/CT scan results. A single 3DCRT plan using the planning target volume is derived from the CT scan only.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIA/IIB or stage IIIA/IIIB disease
* Planning to undergo radiotherapy
* Local or regional nodal recurrence after surgery allowed
* No malignant pleural effusion

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent neoadjuvant and/or concurrent chemotherapy allowed
* No concurrent intensity-modulated radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-02; Primary Completion 2010-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The impact of positron emission tomography (PET)/CT fusion planning on GTV (cm³) vs. planning with CT scan alone | Two treatment plans are centrally reviewed to determine the difference in gross tumor volume between the plans
The impact of positron emission tomography (PET)/CT fusion planning on number of contoured lymph nodes vs. planning with CT scan alone | Two treatment plans are centrally reviewed to determine the difference in number of contoured lymph nodes between the plans
The impact of positron emission tomography (PET)/CT fusion planning on location of involved lymph nodes vs planning with CT scan alone | Two treatment plans are centrally reviewed to determine the difference in location of involved lymph nodes between the plans
The impact of positron emission tomography (PET)/CT fusion planning on lung V20 vs planning with CT scan alone | Two treatment plans are centrally reviewed to determine the difference in lung V20 between the plans
The impact of positron emission tomography (PET)/CT fusion planning vs planning with CT scan alone on mean esophagus dose | Two treatment plans are centrally reviewed to determine the difference in mean esophagus dose between the plans

SECONDARY OUTCOMES:
Rate of elective nodal failures as assessed by failure in previously uninvolved regional lymph nodes at 2 years | From registration to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bradley, MD, Principal Investigator — Mallinckrodt Institute of Radiology at Washington University Medical Center; Jacqueline Brunetti, MD, Study Chair — Sister Patricia Lynch Regional Cancer Center at Holy Name Hospital
Locations (4):
- United States (3):
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - Saint Louis, St Louis, Missouri
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
- McGill Cancer Centre at McGill University, Montreal, Canada

REFERENCES:
- [Result] Bradley J, Bae K, Choi N, Forster K, Siegel BA, Brunetti J, Purdy J, Faria S, Vu T, Thorstad W, Choy H. A phase II comparative study of gross tumor volume definition with or without PET/CT fusion in dosimetric planning for non-small-cell lung cancer (NSCLC): primary analysis of Radiation Therapy Oncology Group (RTOG) 0515. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):435-41.e1. doi: 10.1016/j.ijrobp.2010.09.033. Epub 2010 Nov 13. PMID 21075551